CLINICAL TRIAL: NCT03851692
Title: Intravenous Cannulation In Children During Sevoflurane Induction: Which Time is Adequate
Brief Title: Intravenous Cannulation In Children During Sevoflurane Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Fattouma Bourguiba (Other)
Responsible Party: Principal Investigator, Ben ALI Manel, Clinical Professor, University Hospital Fattouma Bourguiba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0925-0586
Record Dates: First submitted 2018-10-27; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Intravenous Cannulation; Sevoflurane Induction; Child
Keywords: Sevoflurane; Intravenous Cannulation; anesthesia; child
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Intervention Model Description: Prospective randomized single blinded parallel group controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60s (group E) (Active Comparator): Intravenous cannulation was released either 60 s following loss of lid reflex in group E
  Interventions: Other: Intravenous Cannulation (iv placement)
- 90 or 120 s (groupe L) (Active Comparator): Intravenous cannulation was released either 90 or 120 s following loss of lid reflex in group L
  Interventions: Other: Intravenous Cannulation (iv placement)

INTERVENTIONS:
Other: Intravenous Cannulation (iv placement) — The aim of our study is to determine whether one should make intravenous attempts placement during the early induction period (at 60seconds) or lately (90 or 120 s) and waiting until the child receives additional sevoflurane inhalation anesthesia.

SUMMARY:
The early placement of an intravenous (iv) line in children anesthetized with halothane has been shown safe and acceptable compared with later placement. However, there's not well known with sevoflurane use (2). The aim of the investigator's study is to determine whether one should make iv attempts during the early induction period (at 60seconds) or lately (90 or 120 s) and waiting until the child receives additional sevoflurane inhalation anesthesia

DETAILED DESCRIPTION:
the investigators conducted a prospective randomized study, after obtaining Institutional review board approval, which didn't require written parental consent. Children age 1-12 years, undergoing elective general anesthesia via an inhalation induction were randomized to one of three groups of 30 patients each one, for iv placement, either 60s (group E), 90 or 120 s (group L) following loss of lid reflex. Movement on iv placement and incidence of laryngospasm were determined. Difficulty with iv placement was also recorded. Statistical analysis included contingency testing, ANOVA, and non parametric testing. A P-value <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II
* Age from 1 to 12 years old
* Ambulatory surgery under general anesthesia.

Exclusion Criteria:

* Age <1 year or> 12 years
* non-ambulatory surgery,
* contraindication for induction with sevoflurane

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Movement on iv placement | In the first 5 min after the anesthesic induction with sevoflurane
  Number of children who presented movement on iv placement
laryngospasm | Time From Intravenous Cannulation to patient extubation
  The incidence of laryngospasm

CONTACTS AND LOCATIONS:
Overall Officials: Manel Ben Ali, MD, Principal Investigator — University Hospital of Fattouma Bourguiba Monastir TUNISIA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hasan AK, Sivasankar R, Nair SG, Hasan WU, Latif Z. Optimum time for intravenous cannulation after induction with sevoflurane, oxygen, and nitrous oxide in children without any premedication. Paediatr Anaesth. 2018 Feb;28(2):179-183. doi: 10.1111/pan.13308. Epub 2018 Jan 8. PMID 29316032
- [Background] Kumar KR, Sinha R, Chandiran R, Pandey RK, Darlong V, Chandralekha. Evaluation of optimum time for intravenous cannulation after sevoflurane induction of anesthesia in different pediatric age groups. J Anaesthesiol Clin Pharmacol. 2017 Jul-Sep;33(3):371-374. doi: 10.4103/joacp.JOACP_58_16. PMID 29109638